CLINICAL TRIAL: NCT02181400
Title: Pilot Study of Near Infrared Photobiomodulation Treatment for Diabetic Macular Oedema
Brief Title: Near Infrared Photobiomodulation Treatment for Diabetic Macular Oedema
Acronym: NIRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIRD
Record Dates: First submitted 2014-06-27; First posted 2014-07-03 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-01

CONDITIONS: Diabetic Macular Oedema
Keywords: diabetic retinopathy; diabetic macular edema; diabetic macular oedema; near infrared light therapy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- NIR Laser Treatment 25 miiliwatts (mW)/cm2 dose (Active Comparator): The Ellex Integre NIR (near Infrared Light) Laser dose of 25 milliwats(mW)/cm2 for 90 seconds for 12 treatments at 2 to 3 day intervals over 5 weeks.
  Interventions: Device: Ellex Integre NIR laser
- NIR laser treatment 100mW/cm2 dose (Active Comparator): The Ellex Integre NIR Laser dose of 100 mW/cm2 for 90 seconds for 12 treatments at 2 to 3 day intervals over 5 weeks.
  Interventions: Device: Ellex Integre NIR laser
- NIR laser treatment 200mW/cm2 dose (Active Comparator): The Ellex Integre NIR (near Infrared Light) Laser dose of 200 mW/cm2 for 90 seconds for 12 treatments at 2 to 3 day intervals over 5 weeks.
  Interventions: Device: Ellex Integre NIR laser

INTERVENTIONS:
Device: Ellex Integre NIR laser — Each NIR light treatment will consist of a 90 second exposure of the macula of the study eye to the Ellex Integre NIR laser with the patient fixating on the central aiming beam. The laser light beam is 4.5mm in diameter with a central masked area of 1.0 mm diameter containing the central fixation target. In this way the central macula will be spared in the event of an adverse effect of the laser, which we do not anticipate.
  The patient will be seated at the slit lamp laser delivery system and after the eye has been dilated and anesthetised with topical eye drops a standard fundus contact lens will be placed on the eye through which the post area pole will be visualised while the treatment is delivered. There will be 12 treatments administered over a 5 week period.

SUMMARY:
This pilot study aims to establish that treatment with near infrared light (NIR) reduces diabetic macular oedema in patients suffering diabetic retinopathy by exerting a positive beneficial effect at retinal cellular level.

DETAILED DESCRIPTION:
This pilot study aims to establish that treatment with near infrared light (NIR) reduces diabetic macular oedema in patients suffering diabetic retinopathy by exerting a positive beneficial effect at retinal cellular level.

Diabetic retinopathy is a common cause of severe loss of vision and the most common cause of blindness in individuals between the ages of 20 and 65 years in developed countries.Swelling of the central retina or "macular oedema". Patients will be treated in an office clinic,three times a week for a treatment duration of 2 minutes per session, a total of 12 times over the duration of 4 weeks and will be assessed at 8 weeks to establish any change induced in retinal oedema. Safety follow up will be assessed at 3 and 6 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetic Macular Oedema with centre involving thickness of >300µm
2. Age >= 18 years
3. Diagnosis of diabetes mellitus
4. Best corrected visual acuity of 6/9 to 6/60 (letters 77- 33)
5. Intraocular pressure 6 to 25 mmHg
6. Written informed consent has been obtained.

Exclusion Criteria:a) Known allergy to agents used in the study eg. fluorescein b) Women who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using reliable means of contraception. A woman is considered of childbearing potential unless she is postmenopausal and without menses for 12 months or is surgically sterilised c) Loss of vision due to other causes (e.g. age related macular degeneration, myopic macular degeneration, retinal vein occlusion) d) Macular oedema due to other causes e) An ocular condition that would prevent visual acuity improvement despite resolution of oedema (such as foveal atrophy or substantial premacular fibrosis) f) Treatment with intravitreal triamcinolone acetonide (IVTA) within the last 6 months or peribulbar triamcinolone within the last 3 months, or anti vascular endothelial growth factor (VEGF) drugs: ranibizumab and aflibercept, within the last 2 months.

g) Cataract surgery within the last 3 months h) Retinal laser treatment within the last 4 months i) Media opacity including cataract that already precludes adequate macular photography or cataract that is likely to require surgery within 6 months j) Intercurrent severe disease such as septicaemia, any condition which would affect follow-up or photographic documentation (e.g. geographical, psycho-social) k) History of chronic renal failure requiring dialysis or renal transplant l) Blood pressure >180/100 m) Patient has a condition or is in a situation that in the investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-04-19 (Actual); Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark C Gillies, MD PhD, Principal Investigator — Sydney University
Locations (1):
- Sydney Eye Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Derived] Shen W, Teo KYC, Wood JPM, Vaze A, Chidlow G, Ao J, Lee SR, Yam MX, Cornish EE, Fraser-Bell S, Casson RJ, Gillies MC. Preclinical and clinical studies of photobiomodulation therapy for macular oedema. Diabetologia. 2020 Sep;63(9):1900-1915. doi: 10.1007/s00125-020-05189-2. Epub 2020 Jul 14. PMID 32661752

RESULTS

PARTICIPANT FLOW:
Groups:
- NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose: The Ellex Integre NIR (near Infrared Light) Laser dose of 25 milliwats(mW)/cm2 for 90 seconds for 12 treatments at 2 to 3 day intervals over 5 weeks.
  Ellex Integre NIR laser: Each NIR light treatment will consist of a 90 second exposure of the macula of the study eye to the Ellex Integre NIR laser with the patient fixating on the central aiming beam. The laser light beam is 4.5mm in diameter with a central masked area of 1.0 mm diameter containing the central fixation target. In this way the central macula will be spared in the event of an adverse effect of the laser, which we do not anticipate.
  The patient will be seated at the slit lamp laser delivery system and after the eye has been dilated and anesthetised with topical eye drops a standard fundus contact lens will be placed on the eye through which the post area pole will be visualised while the treatment is delivered. There will be 12 treatments administered over a 5 week period.
- NIR Laser Treatment 100mW/cm2 Dose: The Ellex Integre NIR Laser dose of 100 mW/cm2 for 90 seconds for 12 treatments at 2 to 3 day intervals over 5 weeks.
  Ellex Integre NIR laser: Each NIR light treatment will consist of a 90 second exposure of the macula of the study eye to the Ellex Integre NIR laser with the patient fixating on the central aiming beam. The laser light beam is 4.5mm in diameter with a central masked area of 1.0 mm diameter containing the central fixation target. In this way the central macula will be spared in the event of an adverse effect of the laser, which we do not anticipate.
  The patient will be seated at the slit lamp laser delivery system and after the eye has been dilated and anesthetised with topical eye drops a standard fundus contact lens will be placed on the eye through which the post area pole will be visualised while the treatment is delivered. There will be 12 treatments administered over a 5 week period.
- NIR Laser Treatment 200mW/cm2 Dose: The Ellex Integre NIR (near Infrared Light) Laser dose of 200 mW/cm2 for 90 seconds for 12 treatments at 2 to 3 day intervals over 5 weeks.
  Ellex Integre NIR laser: Each NIR light treatment will consist of a 90 second exposure of the macula of the study eye to the Ellex Integre NIR laser with the patient fixating on the central aiming beam. The laser light beam is 4.5mm in diameter with a central masked area of 1.0 mm diameter containing the central fixation target. In this way the central macula will be spared in the event of an adverse effect of the laser, which we do not anticipate.
  The patient will be seated at the slit lamp laser delivery system and after the eye has been dilated and anesthetised with topical eye drops a standard fundus contact lens will be placed on the eye through which the post area pole will be visualised while the treatment is delivered. There will be 12 treatments administered over a 5 week period.
Period: Overall Study
Arm/Group | NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose | NIR Laser Treatment 100mW/cm2 Dose | NIR Laser Treatment 200mW/cm2 Dose
Started | 7 | 7 | 7
Completed | 7 | 7 | 7
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose | NIR Laser Treatment 100mW/cm2 Dose | NIR Laser Treatment 200mW/cm2 Dose | Total
Number analyzed (Participants) | 7 | 7 | 7 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 6 | 10
  >=65 years | 6 | 4 | 1 | 11
Age, Continuous [Mean (Full Range); unit: years] | 73 [67 to 88] | 63 [61 to 88] | 60 [53 to 65] | 65 [53 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 2
  Male | 6 | 6 | 7 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 7 | 7 | 7 | 21
Visual Acuity change [Mean (Standard Deviation); unit: letters] | 64.6 (10.8) | 64.3 (7.3) | 68.8 (13.3) | 65.9 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Change in Measurement in Central Macular Thickness Measured by Spectral Domain Optical Coherence Tomography( OCT) at One Month
Description: Change in measurement( in microns) in central macular thickness as measured by Spectral Domain Optical Coherence Tomography( OCT)
Time Frame: Change from baseline in central macular thickness at one month
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose | NIR Laser Treatment 100mW/cm2 Dose | NIR Laser Treatment 200mW/cm2 Dose
Number analyzed (Participants) | 7 | 7 | 7
micrometers | -25.2 (35.1) | -29.9 (38.6) | -58.9 (45.5)
Statistical Analysis 1: Comparison: NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose vs NIR Laser Treatment 100mW/cm2 Dose vs NIR Laser Treatment 200mW/cm2 Dose; Test type: Other; p = 0.04, ANCOVA

2. Primary Outcome: Change in Measurement in Central Macular Thickness Measured by Spectral Domain Optical Coherence Tomography (OCT) at Two Months
Description: Change in measurement (in microns) in central macular thickness as measured by Spectral Domain Optical Coherence Tomography (OCT)
Time Frame: Change from baseline central macular thickness at two months
Measure: Mean (Standard Deviation); unit: micrometers
Arm/Group | NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose | NIR Laser Treatment 100mW/cm2 Dose | NIR Laser Treatment 200mW/cm2 Dose
Number analyzed (Participants) | 7 | 7 | 7
micrometers | -52.5 (23.6) | -128.6 (51.4) | -114 (59.5)
Statistical Analysis 1: Comparison: NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose vs NIR Laser Treatment 100mW/cm2 Dose vs NIR Laser Treatment 200mW/cm2 Dose; Test type: Other; p = 0.04, ANCOVA

3. Primary Outcome: Change in Total Macular Volume as Measured by Spectral Domain Optical Coherence Tomography at One Month.
Description: The change in total macular volume was taken as the difference between the total macular volume as measured by Spectral Domain Optical Coherence Tomography at 1 month and the total macular volume at baseline
Time Frame: Change from baseline total macular volume at one month
Measure: Mean (Standard Deviation); unit: millimeter cube
Arm/Group | NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose | NIR Laser Treatment 100mW/cm2 Dose | NIR Laser Treatment 200mW/cm2 Dose
Number analyzed (Participants) | 7 | 7 | 7
millimeter cube | 0.1 (0.4) | 0 (0.1) | -0.3 (0.4)
Statistical Analysis 1: Comparison: NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose vs NIR Laser Treatment 100mW/cm2 Dose vs NIR Laser Treatment 200mW/cm2 Dose; Test type: Other; p = 0.12, ANCOVA

4. Primary Outcome: Change in Total Macular Volume as Measured by Spectral Domain Optical Coherence Tomography at Two Months.
Description: The change in total macular volume was taken as the difference between the total macular volume as measured by Spectral Domain Optical Coherence Tomography at 2 month and the total macular volume at baseline
Time Frame: Change from baseline total macular volume as measured by OCT at two months
Measure: Mean (Standard Deviation); unit: millimeters cube
Arm/Group | NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose | NIR Laser Treatment 100mW/cm2 Dose | NIR Laser Treatment 200mW/cm2 Dose
Number analyzed (Participants) | 7 | 7 | 7
millimeters cube | -0.2 (0.1) | 0.2 (0.7) | -0.2 (1.2)
Statistical Analysis 1: Comparison: NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose vs NIR Laser Treatment 100mW/cm2 Dose vs NIR Laser Treatment 200mW/cm2 Dose; Test type: Other; p = 0.32, ANCOVA

5. Secondary Outcome: Change in Logmar Best Corrected Visual Acuity (BCVA) at One Month.
Description: Change in Logmar Best corrected visual acuity (BCVA) from 1 month to that measured at baseline
Time Frame: Change from baseline BCVA measured at one month
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose | NIR Laser Treatment 100mW/cm2 Dose | NIR Laser Treatment 200mW/cm2 Dose
Number analyzed (Participants) | 7 | 7 | 7
letters | 4 (2.0) | 2 (4) | 6 (13)
Statistical Analysis 1: Comparison: NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose vs NIR Laser Treatment 100mW/cm2 Dose vs NIR Laser Treatment 200mW/cm2 Dose; Test type: Other; p = 0.02, ANCOVA

6. Secondary Outcome: Change in Logmar Best Corrected Visual Acuity (BCVA) at Two Months
Description: Change in Logmar Best corrected visual acuity (BCVA) from 2 month to that measured at baseline
Time Frame: Change from baseline BCVA measured at two months
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose | NIR Laser Treatment 100mW/cm2 Dose | NIR Laser Treatment 200mW/cm2 Dose
Number analyzed (Participants) | 7 | 7 | 7
letters | 4 (6) | -2 (7) | -3 (9.5)
Statistical Analysis 1: Comparison: NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose vs NIR Laser Treatment 100mW/cm2 Dose vs NIR Laser Treatment 200mW/cm2 Dose; Test type: Other; p = 0.49, ANCOVA

ADVERSE EVENTS:
Time Frame: AEs and SAEs ocular and non-ocular were reported for the whole period in which the participant was in the trial. 16 weeks
Arm/Group | NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose | NIR Laser Treatment 100mW/cm2 Dose | NIR Laser Treatment 200mW/cm2 Dose
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 7/7 | 4/7 | 6/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NIR Laser Treatment 25 Miiliwatts (mW)/cm2 Dose (N=7) | NIR Laser Treatment 100mW/cm2 Dose (N=7) | NIR Laser Treatment 200mW/cm2 Dose (N=7)
Unrelated to study treatment systemic adverse events (General disorders) | 7 | 4 | 6 — see AE table if needed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/00/NCT02181400/Prot_000.pdf